CLINICAL TRIAL: NCT01281566
Title: Double-blind, Randomized, Placebo-controlled Clinical Trial to Assess the Efficacy and Safety of R051619 (Cisapride Oral Suspension 0.2mg/kg q.i.d) for the Treatment of Feeding Intolerance in Premature Infants
Brief Title: A Study of Cisapride in Premature Infants With Feeding Problems
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor request
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Protfolio/CDT Leader, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR003955; CIS-INT-28
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Infant, Premature; Infant, Newborn
Keywords: Cisapride (Prepulsid); Feeding intolerance; Enteral feeding; Nasogastric tube; Neonate
MeSH Terms: conditions — Premature Birth | interventions — Cisapride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): Cisapride 0.2 mg/kg liquid suspension 4 times a day (q.i.d.) for up to 42 days
  Interventions: Drug: Cisapride
- 002 (Placebo Comparator): Placebo liquid suspension identical in appearance to Cisapride 4 times a day (q.i.d.) for up to 42 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — liquid suspension identical in appearance to Cisapride 4 times a day (q.i.d.) for up to 42 days
  Arms: 002
Drug: Cisapride — 0.2 mg/kg liquid suspension 4 times a day (q.i.d.) for up to 42 days
  Arms: 001

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Cisapride in improving feeding problems in premature newborn infants.

DETAILED DESCRIPTION:
This is a double-blind study where the identity of the treatment assigned (Cisapride or placebo) will not be known to the patient's legal guardian or any study staff involved with the study. Patients will be randomized (assigned by chance) to receive either the drug Cisapride or a placebo (a placebo is identical in appearance to Cisapride but does not contain Cisapride or any active drug) to see if Cisapride is effective in improving feeding problems (referred to as feeding intolerance) in premature newborn infants who cannot tolerate oral feeding by mouth or through a tube going directly to the stomach or intestine. Patients will be given either cisapride at a dose of 0.2 mg/kg or placebo as a liquid suspension through a tube from the nose to the stomach (referred to as a nasogastric tube) 15 minutes before feeding once every 6 hours (or 4 times a day referred to as a q.i.d. schedule).

ELIGIBILITY:
Inclusion Criteria:

* Must be hospitalized and on continuous cardiac monitoring for the duration of the study
* Patient has demonstrated feeding intolerance as defined by the protocol
* Patient's parent or legal guardian must sign the informed consent form

Exclusion Criteria:

* Currently active significant cardiovascular disease, as determined by the neonatologist/physician, including congenital heart disease and heart block (patent ductus arteriosus without cardiac compromise at the time of randomization is acceptable)

Ages: 36 Weeks to 99 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2003-03; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Time from start of study medication to full enteral feeding | Up to 42 days

SECONDARY OUTCOMES:
Number and type of adverse events | Up to 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.